CLINICAL TRIAL: NCT06197061
Title: Comparison of Robot-assisted With Laparoscopic-assisted Modified Soave With Short Muscular Cuff Anastomosis for Classical Hirschsprung Disease
Brief Title: Comparison of Robot-assisted With Laparoscopic-assisted Modified Soave Procedure for Classical Hirschsprung Disease
Acronym: RAMS vs LAMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zunyi Medical College (Other)
Responsible Party: Principal Investigator, zebing Zheng, prof, Zunyi Medical College
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: robot Soave procedure; 82060100 (Other Grant/Funding Number: National Natural Science Foundation of China); ZK-2021-361 (Other Grant/Funding Number: Basic Research Project of Guizhou Province China)
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Hirschsprung Disease
Keywords: Hirschsprung disease; robotic surgery; modified Soave; muscular cuff; Postoperative complications; Efficacy
MeSH Terms: conditions — Hirschsprung Disease; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot-assisted modified Soave group (Experimental): The robotic arms were oriented from the caudal direction. Dissection was begun circumferentially at 1.0 cm above the peritoneal reflection. The rectum was mobilized outside the longitudinal muscle layer, with the anatomical plane farther away from Denonvillier's fascia and the nerve plexus anterior or lateral to the rectum. The mobilization of the rectum reached 4-7 cm into the pelvis. After the robot was unlocked, a circular incision was made 0.5-1 cm from the dentate line, dividing the mucosa upward by 0.5-1.0 cm, breaking through the muscular cuff, and exposing the robotic dissection plane in the pelvis. The diseased colon was then gently pulled out through the anus. The posterior wall of the muscular cuff was completely removed along the left and right sides, accounting for two-thirds of the whole circular muscular cuff to 0.5 cm of the dentate line edge. One third of the anterior wall of the muscular cuff was retained,we then performed Soave's anastomosis.
  Interventions: Procedure: RAMS
- laparoscopic-assisted modified Soave group (Active Comparator): The mesentery of the colon was separated by laparoscopy with the vessel of the pull-through bowel preserved. Under the rectal peritoneal reflex, close to the rectal wall separate with the electric hook, the anterior wall of the rectum was separated to the bladder neck or the posterior wall of the vagina. The posterior wall of the rectum can be separated down to 1cm above the dentate line .a circular incision was made 0.5-1 cm from the dentate line, dividing the mucosa upward by 0.5-1.0 cm, breaking through the muscular cuff, and exposing the robotic dissection plane in the pelvis. The diseased colon was then gently pulled out through the anus. The posterior wall of the muscular cuff was completely removed along the left and right sides, accounting for two-thirds of the whole circular muscular cuff to 0.5 cm of the dentate line edge. One third of the anterior wall of the muscular cuff was retained,we then performed Soave's anastomosis with interrupted 5-0 or 4-0 absorbable sutures.
  Interventions: Procedure: LAMS

INTERVENTIONS:
Procedure: RAMS — The robotic arms were oriented from the caudal direction. Dissection was begun circumferentially at 1.0 cm above the peritoneal reflection. The rectum was mobilized outside the longitudinal muscle layer, with the anatomical plane farther away from Denonvillier's fascia and the nerve plexus anterior or lateral to the rectum. The mobilization of the rectum reached 4-7 cm into the pelvis. After the robot was unlocked, a circular incision was made 0.5-1 cm from the dentate line, dividing the mucosa upward by 0.5-1.0 cm, breaking through the muscular cuff, and exposing the robotic dissection plane in the pelvis. The diseased colon was then gently pulled out through the anus. The posterior wall of the muscular cuff was completely removed along the left and right sides, accounting for two-thirds of the whole circular muscular cuff to 0.5 cm of the dentate line edge. One third of the anterior wall of the muscular cuff was retained,we then performed Soave's anastomosis.
  Arms: Robot-assisted modified Soave group
Procedure: LAMS — The mesentery of the colon was separated by laparoscopy with the vessel of the pull-through bowel preserved. Under the rectal peritoneal reflex, close to the rectal wall separate with the electric hook, the anterior wall of the rectum was separated to the bladder neck or the posterior wall of the vagina. The posterior wall of the rectum can be separated down to 1cm above the dentate line. After the laparoscopy was unlocked, a circular incision was made 0.5-1 cm from the dentate line, dividing the mucosa upward by 0.5-1.0 cm, breaking through the muscular cuff, and exposing the laparoscopic dissection plane in the pelvis. The diseased colon was then gently pulled out through the anus. The posterior wall of the muscular cuff was completely removed along the left and right sides, accounting for two-thirds of the whole circular muscular cuff to 0.5 cm of the dentate line edge. One third of the anterior wall of the muscular cuff was retained,we then performed Soave's anastomosis.
  Arms: laparoscopic-assisted modified Soave group

SUMMARY:
Hirschsprung disease (HSCR) is a rare congenital intestinal disease characterized by the absence of ganglion cells in the distal rectum, extending for variable distances into the proximal intestine.The "pull-through" reconstruction procedure described in 1949 by Orvar Swenson involving the removal of the aganglionic bowel and creating an anastomosis between the normally innervated bowel and the anal canal, remains the standard surgical approach for HSCR today. However, as rectal dissection by laparotomy in infants is technically difficult and can result in high rates of complications, other pull-through techniques were developed and several techniques are still widely used today.

In our institute, we developed the laparoscopic-assisted modified Soave with short muscular cuff anastomosis in July 2017, and achieved good therapeutic effects. However, there have some patients suffered soiling incidents in the short period post-surgery.

Therefore, we developed the robot-assisted modified Soave with short muscular cuff anastomosis procedures to protect the vital nerve and blood vessels of the pelvis from injury, decrease the injury of the sphincter.

this clinical trials was to compare the efficacy of robot-assisted and laparoscopic-assisted modified Soave with short muscular cuff anastomosis procedures for classical Hirschsprung disease (HSCR).

DETAILED DESCRIPTION:
Soave's first report on the endorectal pull-through without anastomosis approach to the treatment of Hirschsprung disease (HSCR) dates back to 1963. With the rapid development of laparoscopic operations in the early 1990s, Georgeson et al reported a technique utilizing laparoscopic dissection of the rectum combined with anal mucosal dissection in 1995. Subsequently, many laparoscopic approaches to modified Soave-Georgeson procedures were described, including short muscular cuff anastomosis, long cuff dissection, and short V-shaped partially resected cuff anastomosis.The purpose of these modifications is to decrease postoperative complications due to internal anal sphincter achalasia and rectal cuff.

Wester et al used a short cuff operation that retained a muscular cuff of 1-2 cm and achieved excellent outcomes. Due to our increased experience to Soave-Georgeson operation, we have modified the Soave-Georgeson procedure that developed laparoscopic stepwise gradient cutting muscular cuff procedure and shortened the muscular cuff to approximately 1-2 cm in neonates and infants, or 3-4 cm in children. Good results using the laparoscopic stepwise gradient cutting muscular cuff (LSGC) procedure have been reported by Zheng et al.

Although a few patients suffered enterocolitis of the LSGC procedure, we found that the incidence of enterocolitis in patients with a 1-2cm muscular cuff was lower than that in patients with a 3-4 cm muscular cuff. According to the above finding, we developed the laparoscopic-assisted modified Soave with short muscular cuff anastomosis in July 2017, and achieved good therapeutic effects. However, there have some patients suffered soiling incidents in the short period post-surgery.

Therefore, we developed the robot-assisted modified Soave with short muscular cuff anastomosis procedures to protect the vital nerve and blood vessels of the pelvis from injury, decrease the injury of the sphincter.

this clinical trials was to compare the efficacy of robot-assisted and laparoscopic-assisted modified Soave with short muscular cuff anastomosis procedures for classical Hirschsprung disease (HSCR).

ELIGIBILITY:
Inclusion Criteria:

* 1.Age no more than 18 years 2.Hirschsprung disease diagnosed by biopsy 3.Performed modified Soave procedure for treatment.

Exclusion Criteria:

* 1.Total colonic aganglionosis 2.Descending/transverse colon Hirschsprung disease 3.Combined with Down syndrome 4.preoperative enterostomy 5.refused to participate

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-02-07 (Actual); Primary Completion 2024-02-08 (Estimated); Study Completion 2024-10-10 (Estimated)

PRIMARY OUTCOMES:
Soiling | 2 years
  The incidence of complication of Soiling between two groups.
Enterocolitis | 2 years
  The incidence of complication of enterocolitis between two groups.

SECONDARY OUTCOMES:
operative time | 2 years
  The operative time(minute) were analysis in two groups
The anal dissection time | 2 years
  The anal dissection time(minute) were analysis in two groups
length of hospitalization | 2 years
  The postoperative length of hospitalization (days) were analysis between two groups
blood loss | 2 years
  The Blood loss were analysis in two groups
Perianal dermatitis | 2 years
  The incidence of complication of Perianal dermatitis between two groups
Urinary incontinence | 2 years
  The incidence of complication of Urinary incontinence between two groups
Anastomotic leakage | 2 years
  The incidence of complication of Anastomotic leakage between two groups
Cuff abscess | 2 years
  The incidence of complication of Cuff abscess between two groups
Anastomotic strictures | 2 years
  The incidence of complication of Anastomotic strictures between two groups
Sphincter spasm | 2 years
  The incidence of complication of Sphincter spasm between two groups
Staining | 2 years
  The incidence of complication of Staining between two groups
Constipation | 2 years
  The incidence of complication of Constipation between two groups
bowel function score (BFS) | 4 years
  Children aged ≥ 4 years were assessed twice for each score. A BFS ≥ 17 was represented as the lower limit of good/normal functional outcomes as more than 90% of people aged ≥ 4 years in the normal population met this criterion
postoperative fecal continence (POFC) score | 4years
  postoperative fecal continence (POFC) score focused on SNS-related incontinence

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Miyano G, Koga H, Okawada M, Doi T, Sueyoshi R, Nakamura H, Seo S, Ochi T, Yamada S, Imaizumi T, Lane GJ, Okazaki T, Urao M, Yamataka A. Rectal mucosal dissection commencing directly on the anorectal line versus commencing above the dentate line in laparoscopy-assisted transanal pull-through for Hirschsprung's disease: Prospective medium-term follow-up. J Pediatr Surg. 2015 Dec;50(12):2041-3. doi: 10.1016/j.jpedsurg.2015.08.022. Epub 2015 Aug 28. PMID 26386879
- [Result] Neuvonen MI, Kyrklund K, Rintala RJ, Pakarinen MP. Bowel Function and Quality of Life After Transanal Endorectal Pull-through for Hirschsprung Disease: Controlled Outcomes up to Adulthood. Ann Surg. 2017 Mar;265(3):622-629. doi: 10.1097/SLA.0000000000001695. PMID 28169931
- [Result] Crippa J, Grass F, Dozois EJ, Mathis KL, Merchea A, Colibaseanu DT, Kelley SR, Larson DW. Robotic Surgery for Rectal Cancer Provides Advantageous Outcomes Over Laparoscopic Approach: Results From a Large Retrospective Cohort. Ann Surg. 2021 Dec 1;274(6):e1218-e1222. doi: 10.1097/SLA.0000000000003805. PMID 32068552
- [Result] Zhang MX, Zhang X, Chang XP, Zeng JX, Bian HQ, Cao GQ, Li S, Chi SQ, Zhou Y, Rong LY, Wan L, Tang ST. Robotic-assisted proctosigmoidectomy for Hirschsprung's disease: A multicenter prospective study. World J Gastroenterol. 2023 Jun 21;29(23):3715-3732. doi: 10.3748/wjg.v29.i23.3715. PMID 37398887